CLINICAL TRIAL: NCT05419297
Title: True Functional Restoration and Analgesia in Non-Radicular Low Back Pain: a Prospective, Double Blind, Placebo-controlled Study of Buccal Buprenorphine
Brief Title: True Functional Restoration and Analgesia in Non-Radicular Low Back Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carolinas Pain Institute (Other)
Collaborators: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIR CLBP 8.16.21
Record Dates: First submitted 2021-12-08; First posted 2022-06-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Back Pain Lower Back Chronic; Chronic Pain
Keywords: pain
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: A double blind, placebo controlled, phase IV clinical trial. Following a two week washout of opioid medication, a two week single blind placebo lead in, subjects will be randomized into two groups. One group to receive placebo film, and the other to be titrated to effect with buprenorphine buccal film.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Two designated staff will be unblinded, and be responsible for providing the subjects with envelopes containing either drug or placebo. Principal investigator and the remainder of the staff will be blinded throughout the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active drug arm (Active Comparator): Subjects who meet eligibility criteria and complete a single blind placebo lead in will be provided placebo buprenorphine buccal film that mimics the actual drug comparator and is continued by a blinded individual throughout the duration of the trial.
  Interventions: Drug: Buprenorphine Buccal Film [Belbuca]; Other: Urine Drug Screening; Device: actigraph; Behavioral: PROMIS 29; Other: sit to stand test; Other: numerical rating scale pain score; Behavioral: patient global impression of function; Behavioral: PROMIS - sleep
- Placebo arm (Placebo Comparator): Subjects who meet eligibility criteria and complete a single blind placebo lead in will be provided active buprenorphine buccal film that is titrated to the effective dose and continued by a blinded individual throughout the duration of the trial.
  Interventions: Other: Urine Drug Screening; Device: actigraph; Behavioral: PROMIS 29; Other: sit to stand test; Other: numerical rating scale pain score; Behavioral: patient global impression of function; Behavioral: PROMIS - sleep

INTERVENTIONS:
Drug: Buprenorphine Buccal Film [Belbuca] — buprenorphine buccal film is indicated for the management of pain severe enough to require daily, around-the-clock, long-term opioid treatment and for which alternative treatment options are inadequate.
  Other Names: Belbuca
  Arms: Active drug arm
Other: Urine Drug Screening — Urine drug screening to include controlled prescription medication as well as illicit substances to monitor compliance
Device: actigraph — Subjects will wear this device to monitor sleep and activity
  Other Names: Garmin
Behavioral: PROMIS 29 — questionnaire will be administered once a week via e-dairy to monitor mood and sleep
Other: sit to stand test — Subjects will complete this daily with specific instructions through the e-diary
Other: numerical rating scale pain score — subjects will be asked a pain score in the morning, prior to, and after sit-to-stand testing, and at night
Behavioral: patient global impression of function — subjects will be asked three questions once a day to assess their personal impression of functional status
Behavioral: PROMIS - sleep — Subjects will answer 5 questions about sleep every morning via e-diary

SUMMARY:
To study the response of objective and quasi-objective 'True' functional outcomes, analgesia and safety in chronic non-radicular back pain to buprenorphine buccal film (BBF) using a small 'n' phase IV design. To assess associations between traditional pain relevant subjective outcomes and objective or quasi-objective functional outcomes; In a small 'n' construct, to assess more powerful, 'new' statistical methods (e.g. hierarchical linear models, joint trajectory analysis) compared to traditional methods, in the context of increased power, more objective outcomes and cost savings.

First a 2-week washout of any opioid medication (if necessary; if not necessary subject can proceed directly to); baseline week (Single Blind Placebo Lead In (SBPLI), using the placebo film resembling the 150mcg dose; then randomization to a ~ 2 week up titration either to effective Buprenorphine Buccal Film (BBF) dose 2 day average pain better than or equal to 3/10 NRS), highest tolerated dose BBF and/or maximum dose BBF of 900 mcg BID, or identical placebo material up to these parameters. This up titration is at the discretion and timing of the blinded and experienced PI. Subject will be allowed two doses of hydrocodone/acetaminophen 5/325 daily during the washout period.

A single experienced practitioner will manage the titration as to safety, detail and timing; and determine when the subject enters the 8 week stable dose trial; this practitioner will remain blinded throughout unless there is an urgent, safety reason for unblinding

DETAILED DESCRIPTION:
Scientific/Medical Rationale:

Improved function is a high yield goal in back pain in specific, and pain in general. There are a number of self-report scales measuring 'physical functioning', 'quality of life' or ability to complete activities of daily living available. Unfortunately these tests, though sometimes mentioned as 'tests of physical function', retain the significant limitation of being fully subjective as they rely entirely on subject perception and report. These subjective metrics are considered useful in that they show good preliminary correlation with measured functional abilities and true functional performance. There have been many attempts to bring more objective and quantitative functional scales to bear, and these efforts have achieved variable success. Scales that are recorded by a professional observer, such as a physical therapist, lend more 'objectivity' to the assessment, as with the Barthel index. The Functional Capacities Evaluation (FCE) type metrics are highly validated, although geared more toward patients with back pain in the forensic arena. As such they are not as yet practical in the context of CLBP research, multi-center trials, or even the clinic.

Subjective, yet quantified pain ratings are commonly used to follow a patient's response to analgesic treatment,and although having good clinical value for within-subject comparison, between-subject contrasts are less reliable. Multiple factors including culture, memory, the meaning and context of pain, personality types, affective state and a variety of operant variables can influence reported pain,making these outcomes less scientifically adequate than more objective outcomes.

Objective and Quasi-objective instruments have been developed to assess some relevant aspects of the pain experience. For instance, gross functional assessments, such as return to work and health care utilization, have been adapted and validated for pain research. While fully objective testing such as fMRI holds the promise of being able to quantify human pain, this will not be practical in the near future. As there will always be a need for simple "bedside" measures and practical pain laboratory testing, as well as a great need to add objectivity to this otherwise subjective diagnostic set. Logically, function should be a high priority outcome in pain research.

Many measures have been validated over the years that can concurrently assess psychological spheres of the pain experience. While it is clear that the impact of pain and mood are critical components for characterizing the overall clinical pain experience, unfortunately the pain literature is based entirely on self-report psychometric scales, and the subjective nature of these measures make them less than fully satisfactory for research. Thus, there is a critical need to shift the paradigm away from subjective measures (where possible) to more objective methodologies. It is likely that objectification will lower cost in clinical trials through the mechanism of improved power (thus lower numbers of subjects required to demonstrate statistical response).

Finally, traditional statistical schemes require large, expensive trials to show significance; the use of more powerful techniques such as hierarchical statistical models with time series analysis and Bayesian analysis will allow for smaller, less expensive trials to be conducted.

Drugs, Dosages, and Regimens:

First a 2-week washout of any opioid medication (if necessary; if not necessary subject can proceed directly to); baseline week (Single Blind Placebo Lead In (SBPLI), using the placebo film resembling the 75 mcg dose; then randomization to a ~ 2 week up titration either to effective Buprenorphine Buccal Film (BBF) dose 2 day average pain better than or equal to 3/10 NRS), highest tolerated dose BBF and/or maximum dose BBF of 900 mcg BID, or identical placebo material up to these parameters. This up titration is at the discretion and timing of the blinded and experienced PI. Subject will be allowed two doses of hydrocodone/acetaminophen 5/325 daily during the washout period.

A single experienced practitioner will manage the titration as to safety, detail and timing; and determine when the subject enters the 8 week stable dose trial; this practitioner will remain blinded throughout unless there is an urgent, safety reason for unblinding.

Patient population:

A total of 36-40 outpatients of age 18-65, any gender or race with Chronic Non-Radicular low Back Pain (≥ 3 months; CNRBP) diagnosed by history and physical examination will be identified for the trial. Subjects will be recruited from outpatient pain management offices.

Materials and instruments:

* Personal Health History Subjects will be asked to complete a Personal Health History Form at their first visit. This general questionnaire will assess demographic information (sex, age, marital status, race/ethnicity, and education), pain history (injury, onset/duration, description, self-reported diagnostic testing history, and treatment history), and general health history (other medical/surgical history, concurrent medications, health behaviors, a general symptom checklist, and health-care utilization).
* Numeric Rating Scale (NRS): the NRS is a convenient, understandable, and accessible quantification of pain that is often used in pain research. It will be used on the e-diary, at phone contacts, at defined moments in functional testing (before and after a function) and in the clinical visits. The use of the metric in any context will always be referenced as "Pain on a zero to ten scale, with zero being no pain and 10 being the worst pain imaginable".
* Pain Disability Index30: A seven-item, validated instrument that assesses perceived disability in seven key life areas. It provides a total disability score, and is an indirect measure of self-efficacy that will be acquired at all in person visits.
* Patient's Global Impression of Function The PGIF is a 10 point scale (0= no functional limitation, 10= non-functional) and asks the subject to rate his/her Function and Activities of Daily Living.
* PROMIS-29 The P-29 is a distillation of multiple psychometric scores using Item Response Theory.
* Functional Testing Protocol ©: Quasi-objective measures of functional abilities will be obtained.
* Actigraph (whole body 3d accelerometer type system) Participants will wear this device from the beginning to the end of the trial. The data will provide different indexes of participants' level of activity and activity organization, and these functional parameters will also be measured by other psychometric methods. Activity will be monitored via data portal for compliance by the research staff and PI.

Study Design:

Following wean of opioid medication, if necessary, all subjects will participate in a two week single blind placebo lead in to wash out any placebo response. Following the single blind placebo lead in, subjects will be randomized into either a placebo group, or active drug group. Both groups will be titrated to effect during a two week period. Subsequently, subjects will then participate in a total of 12 visits, some telephone, some in person. Throughout the duration of the study, participants will be asked to fulfill daily e-diary requirements which will include NRS, Patient Global Impression of Function, Patient Global Impression of Sleep, and some subjective functional testing. Subjects will also wear an actigraph device which will provide data about sleep and daily movements. Urine drug screening and pill counts will be completed at all in person visits.

Side effects: Subjects who report intolerable side effects will be released from the study.

Intolerable side effects would be defined as:

• Allergy to the study drug with rash, anaphylaxis, pruritis, respiratory depression, or any other symptom that is deemed by the subject as "intolerable".

Common side effects associated with Buprenorphine Buccal Film include, but are not limited to:

* Nausea
* Vomiting
* Feeling sleepy (sedation)
* Feeling drunk
* Constipation
* Dry mouth
* Muscle weakness
* Headache
* Skin Rash
* Dizziness
* Blurred vision
* Feeling hot
* Flu-like illness
* Bladder spasm
* Low blood pressure
* Respiratory depression (slowed
* breathing)
* Pupil narrowing
* Sweating
* Itching
* Hives
* Bronchospasm (difficulty
* breathing)
* Anaphylactic Shock (severe
* allergic reaction)
* Elevated cerebrospinal fluid
* pressure (which could lead to
* decreased blood flow to the
* brain)

Safety Information/data:

Screen: Subjects will be excluded if hypersensitivity to buprenorphine or Belbuca®, subjects with severe or untreated psychiatric disturbance (e.g. mania, depression [esp suicidality], anxiety, substance dependent), subjects with a clinical diagnosis of spinal stenosis, fibromyalgia or polymyalgia rheumatic, subjects with severe ongoing or unaddressed medical conditions (e.g. Renal or Hepatic disease [creatinine>1.5 ml/dl; AST or ALT> 3x normal limit], Severe or uncontrolled hypertension, pulmonary disease, seizure disorder, gastroparesis or urinary retention.

Each visit: vital signs, medical events, side effects and device and drug compliance will be reviewed; concerns and problems will be solicited.

Phone contacts: side effects and device and drug compliance will be reviewed; concerns and problems will be solicited by open ended questions.

Minor, non-significant side effects or adverse events that occur during the study will be recorded in the subject's chart and on an adverse event reporting form. Any serious adverse events or side effects that occur will be recorded in the subject's chart and on the adverse events reporting form and will be reported immediately to the WCG IRB, the Food and Drug Administration, and BDSI officials. An adverse event will be considered serious if it is fatal or immediately life threatening or requires or prolongs inpatient hospitalization, necessitates long-term outpatient treatment, causes permanent disability, is a congenital anomaly, cancer, or overdose. Questions of 'tolerance' will be considered and decided at the discretion of the PI in the context of these reports in consultation with the subject, and if necessary, with BDSI officials. Serious and unexpected adverse events will be reported to the IRB within 24 hours of discovery.

Data will be continually monitored by the study coordinator and consultant and regularly reported to the principal investigator who will review the data and all adverse events after each subject is studied.

ELIGIBILITY:
Inclusion Criteria:

1. Meets our criteria for CNRBP:

   * Pain of 3 months or more duration
   * non-radiating (below buttocks or above lower back pain)
   * no decreased sensation or allodynia/hyperalgesia in a radicular pattern
   * no reflex asymmetry
   * no frank weakness or atrophy
   * no non-pain sensory or reflex changes
2. If female, not pregnant or breast feeding, and not currently attempting to conceive; if of childbearing potential, use of a highly effective method of birth control (as determined by Pl).
3. Able to read and speak English and provide informed consent.
4. Age 18-65.
5. Able to understand and comply with all data collection methodology, and demonstrated ability to manage the electronic diary system (as tested in 'detox' and baseline/SBPLI period).
6. Subjects may continue any non-opioid stable scheduled drug regimen with no changes during the course of study, hydrocodone/acetaminophen 5/325 up to two doses per day along with Tylenol 2g/day are the only allowed rescue medications. Subjects are asked not to use the rescue medication 12 hours or less before testing.
7. Subjects taking opioids must agree to 'detoxify' for the protocol under the supervision of the study medical personnel. Subjects may use hydrocodone/acetaminophen 5/325 twice daily for breakthrough pain, as provided to them during the study, and must use only the hydrocodone/acetaminophen provided (with a pill count is a secondary outcome)
8. Subjects must agree to try to stay as functional as possible (defined by only tolerable increase in pain with function or function testing)
9. Must have 'average' pain greater than or equal to 4 and no greater that 9 on a 10-point NRS scale at phone screening and first visit
10. Subjects must have and maintain a working phone
11. CMP, CBC, UDS, EKG within normal limits at the discretion of the PI.

    -

Exclusion Criteria:

1. Subjects with hypersensitivity to Opioids, Acetaminophen, buprenorphine or Belbuca®
2. Subjects taking equal to or more than 100 morphine milliequivalents,
3. Subjects with severe or untreated psychiatric disturbance (e.g. mania, depression [esp suicidality], anxiety, substance use disorder etc). This exclusion at the discretion of the PI.
4. A known or admitted history of opioid abuse, diversion or addiction.
5. Subjects with severe, ongoing or unaddressed medical conditions (e.g. Renal or Hepatic disease i. [creatinine>1.5 ml/dl; AST or ALT> 2x normal limit], severe or uncontrolled hypertension, pulmonary ii. disease, seizure disorder or gastroparesis or urinary retention.
6. Subjects with a clinical diagnosis of fibromyalgia, polymyalgia rheumatica, spinal stenosis or non-osteoarthritis i. rheumatologic disease or severe chronic pain disorder of other body regions.
7. Subjects who are currently talking MAO inhibitors (must have been off for > 14 days)
8. Subjects with planned surgery or invasive/interventional procedures.
9. Subjects must be willing to comply with visit and phone contact schedule, and try to stay as active and 'functional' as they can.
10. Subjects cannot be involved in any litigation concerning Workers Compensation or lawsuit concerning injury.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Numberic Rating Scale | 20 weeks
  Numeric rating scale pain scores (0-10; 0- no pain, 10 - worst pain imaginable) will be recorded on a daily basis in the placebo and active comparator groups.
Patient global impression of function | 20 weeks
  2 questions administered through an e-dairy on a daily basis to assess subject's impression fo function. Numeric scale: 0 no functional impairment due to pain; 10 total functional impairment due to pain
Patient Reported Outcomes Information System - Sleep | 20 weeks
  Subjects will be provided a 5 point scale to rate sleep which will be scored. 4 - 20 higher score shows the most sleep disturbance, lower score is no sleep disturbance
Activity - steps per day | 20 weeks
  Actigraph data, using a garmin device, will be gathered to record the number of steps the subject took in a 24 hour time period
Activity - time sitting | 20 weeks
  Actigraph data, using a garmin device. Time sitting in hours and minutes will be recorded on a 24 hour time block
Sit to stand test | 20 weeks
  Function - subjects will perform sit to stand test to measure pain and ability to perform such activity to compare the placebo and active comparator groups.
activity -sleep | 20 weeks
  actigraph data, utilizing a garmin device, will be gathered recording time the subject was sleeping based on movements and heart rate in a 24 hour period
Timed stair climb | 20 weeks
  9 steps will be ascended with or without the use of a handrail. Time will be recorded in seconds.
Patient Reported Outcomes Information System - 29 | 20 weeks
  29 questions about mood, sleep, and function will be gathered on a weekly basis via e-diary. This is scored, with 29 being the best outcome, and 100 the worst

SECONDARY OUTCOMES:
Function | 20 weeks
  Sit to stand and stair climb results will be compared to the patient's subjective report in the patient global impression of function questionairre.
Sleep | 20 weeks
  Patient Reported Outcomes Information System - Sleep score will be compared with the actual sleep data gathered via actigraph
Activity | 20 weeks
  Subject reported numerical rating system score will be compared with number of steps during a 24 hour period gathered via actigraph device.
Bayesian analysis | 20 weeks
  Bayesian analysis will be utilized to determine statistically significant differences in all parameters amongst the two arms as well as subjective and objective data comparisons

CONTACTS AND LOCATIONS:
Overall Officials: AMANDA A ZIMMERMAN, PA-C, Principal Investigator — West Forsyth Pain Management
Locations (1):
- Carolinas Pain Institute, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No